CLINICAL TRIAL: NCT03614325
Title: Virtual Reality in the Operating Room: Using Immersive Relaxation as an Adjunct to Anesthesia
Brief Title: Virtual Reality in the Operating Room
Acronym: OR-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: VRHealth Group Ltd (Industry)
Responsible Party: Principal Investigator, Brian O'Gara, Attending Anesthesiologist, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P000398
Record Dates: First submitted 2018-07-09; First posted 2018-08-03 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia, Intravenous; Pain, Postoperative; Delayed Recovery From Anesthesia; Satisfaction; Relaxation Therapy
MeSH Terms: conditions — Pain, Postoperative; Delayed Emergence from Anesthesia; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Anesthesia Care (No Intervention): Patients in the usual care arm will undergo the current standard of care for hand/wrist surgery and postoperative recovery. They will be asked to refrain from using a virtual reality headset during their surgery.
- Virtual Reality Immersive Relaxation (Experimental): Patients in the experimental group will wear a headset and be immersed in a virtual reality environment during their surgery. There are various short videos and environments such as sitting on a beach that are designed to promote relaxation and calmness.
  Throughout their surgery patients will be monitored according to current anesthesia standards. The relaxation programming will run for the duration of the operative procedure. At the end of the procedure the headset will be removed and standard postoperative care will commence.
  Interventions: Other: Virtual Reality Immersive Relaxation

INTERVENTIONS:
Other: Virtual Reality Immersive Relaxation — The software developed by VRHealth allows patients to select from scenery such as mountains, the beach or from a selection of short videos, which are intended to promote relaxation.
  Arms: Virtual Reality Immersive Relaxation

SUMMARY:
This is a randomized, controlled trial designed to investigate whether the use of virtual reality immersive relaxation during hand/arm operations can allow for a relaxing operating room experience for patients while potentially reducing anesthesia requirements.

DETAILED DESCRIPTION:
The proposed study is a randomized, controlled trial to evaluate the effectiveness of VR as an adjunct to standard anesthetic practice for upper extremity surgery. Patients will be randomized to undergo immersion relaxation via the use of VR during their procedure or control. In both groups patients will undergo regional anesthesia preoperatively according to standard practice. Patients will then be assessed postoperatively to assess the intraoperative propofol dose between groups, as well as secondary outcomes including patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing upper extremity (hand, wrist, arm, and/or elbow) surgery at BIDMC under MAC

Exclusion Criteria:

* Age < 18
* Open wounds or active infection of the face or eye area
* History of seizures or other symptom linked to an epileptic condition
* Patients who plan to wear hearing aids during the procedure
* Patients with a pacemaker or other implanted medical device
* Droplet or airborne precautions (as determined by BIDMC infection control policy)
* Non-English speaking
* Patients who require deep sedation
* Patients who are deemed ineligible to approach by the surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Gara, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faruki A, Nguyen T, Proeschel S, Levy N, Yu J, Ip V, Mueller A, Banner-Goodspeed V, O'Gara B. Virtual reality as an adjunct to anesthesia in the operating room. Trials. 2019 Dec 27;20(1):782. doi: 10.1186/s13063-019-3922-2. PMID 31882015

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Reality Immersive Relaxation: Patients in the experimental group will wear a headset and be immersed in a virtual reality environment during their surgery. There are various short videos and environments such as sitting on a beach that are designed to promote relaxation and calmness.
  Throughout their surgery patients will be monitored according to current anesthesia standards. The relaxation programming will run for the duration of the operative procedure. At the end of the procedure the headset will be removed and standard postoperative care will commence.
  Virtual Reality Immersive Relaxation: The software developed by VRHealth allows patients to select from scenery such as mountains, the beach or from a selection of short videos, which are intended to promote relaxation.
Period: Overall Study
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Started | 20 | 20
Completed Intervention | 17 | 17
Completed | 15 | 16
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Surgery Cancelled | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Surgery never scheduled | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.1) | 48.7 (19.0) | 49.4 (0.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] — BMI - Body Mass Index
  Kg/m^2 | 28.7 (5.2) | 28.1 (4.8) | 28.4 (.12)
Diabetes [Count of Participants; unit: Participants] | 4 | 2 | 6
Hypertension [Count of Participants; unit: Participants] | 6 | 9 | 15
Dyslipidemia [Count of Participants; unit: Participants] | 6 | 5 | 11
Obesity [Count of Participants; unit: Participants] | 7 | 3 | 10
COPD [Count of Participants; unit: Participants] | 4 | 3 | 7
Depression [Count of Participants; unit: Participants] | 6 | 3 | 9
Anxiety [Count of Participants; unit: Participants] | 3 | 2 | 5
Previous Use of VR [Count of Participants; unit: Participants]
  Never | 13 | 10 | 23
  Once | 2 | 3 | 5
  A few times | 1 | 4 | 5
  Many times | 1 | 0 | 1
Procedure Type [Count of Participants; unit: Participants] — Multiple bookings per case are possible
  Participants
    Carpal Tunnel | 4 | 4 | 8
    Dupuytren's contracture | 1 | 2 | 3
    Tendon/ligament repair | 5 | 3 | 8
    Ganglion removal | 3 | 3 | 6
    Ulnar neurolysis/decompression | 2 | 4 | 6
    Mass/cyst excision | 3 | 1 | 4
    Reduction and/or internal fixation | 2 | 3 | 5
    Other | 4 | 2 | 6
Surgery Length [Median (Inter-Quartile Range); unit: minutes] | 27.0 [16.5 to 45.5] | 19.0 [12.5 to 51.0] | 23 [14.5 to 48.25]
Regional Anesthetic [Count of Participants; unit: Participants]
  Supraclavicular | 4 | 7 | 11
  Infraclavicular | 11 | 8 | 19
  None/data missing | 2 | 2 | 4
Regional Anesthetic [Median (Inter-Quartile Range); unit: mg]
  Bupivacaine | 100 [75 to 100] | 100 [67.5 to 100] | 100 [71.25 to 100]
  Mepivacaine | 240 [200 to 300] | 200 [200 to 200] | 220 [200 to 250]
Regional Anesthetic [Count of Participants; unit: Participants] — Number of patients administered Midazolam for anxiolysis during the preoperative nerve block
  Participants | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Propofol Dose
Description: Total propofol dose (mg/kg/min) administered intraoperatively will be measured for the duration of the procedure.
Time Frame: 60 minutes
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
mg/kg/min | 0.14 [0.12 to 0.21] | 0.00 [0.00 to 0.01]

2. Secondary Outcome: Other Intraoperative Anesthetics or Analgesics Administered
Description: Total dose of additional anesthetics (other than propofol) or analgesics administered intraoperatively will be measured for the duration of the procedure.
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
Participants
  Ketamine | 1 | 2
  Fentanyl | 2 | 1
  Ketorolac | 4 | 2
  Supplemental local block | 1 | 7

3. Secondary Outcome: Total Intraoperative Propofol Administered
Description: Total propofol dose (mg bolus, mg infusion, and mg total) administered intraoperatively will be measured for the duration of the procedure.
Time Frame: 60 minutes
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
mg
  Protofol bolus | 50 [0 to 65] | 0 [0 to 20]
  Propofol infusion | 223 [162 to 384] | 0 [0 to 0]
  Propofol total dose | 260 [203 to 469] | 0 [0 to 30]

4. Secondary Outcome: Length of PACU Stay
Description: The length of the patients stay in the Post Anesthesia Care Unit will be measured in minutes
Time Frame: Duration of the patient's stay in the post anesthesia care unit, 100 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
minutes | 75.0 [57.5 to 89.0] | 53.0 [43.0 to 72.0]

5. Secondary Outcome: Pain Assessed by Eleven Point Numerical Rating Scale
Description: Clinically documented pain scores will be recorded on a scale from 0 (best outcome) to 10 (worst outcome).
Time Frame: Duration of stay in the post anesthesia care unit, 100 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
units on a scale | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Overall Patient Satisfaction
Description: Patient satisfaction will be assessed using a survey which asks about ease of use, programming preferences and overall study satisfaction. The satisfaction score will be reported on a scale from 0 (worst outcome; very unsatisfied) to 100 (best outcome; very satisfied).
Time Frame: PACU discharge
Population: Modified intention to treat (those randomized who completed study protocol)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
units on a scale | 100 [100 to 100] | 92 [77 to 100]

7. Secondary Outcome: Patient Survey: Agreement With the Following Statements (0-100)
Description: Patients are asked their level of agreement with statements about how well their pain was controlled, whether they felt anxious, whether they felt relaxed, whether they could remember their time in surgery, and whether they would be interested in using VR for another surgery. The total score will be reported on a scale from 0 (worst outcome, no agreement) to 100 (best outcome, total agreement).
Time Frame: PACU discharge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
units on a scale
  My pain was controlled | 100 [100 to 100] | 100 [76 to 100]
  I felt relaxed | 100 [100 to 100] | 99 [79 to 100]
  I felt anxious | 0 [0 to 2] | 0 [0 to 30]
  I remember being aware of how I felt in the OR | 0 [0 to 0] | 97 [79 to 100]
  I would be interested in VR for future surgery | 100 [68 to 100] | 100 [69 to 100]

8. Secondary Outcome: Hand Disability (QuickDASH)
Description: As assessed by the Quick Disabilities of the Arm, Shoulder, and Hand (DASH) score; a patient reported outcome scale regarding hand disability. Scores range from 0 (no disability) to 100 (most severe disability).
Time Frame: One month postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale, 0 - 100
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
score on a scale, 0 - 100 | 40.9 [27.3 to 59.1] | 20.5 [9.1 to 40.9]

9. Secondary Outcome: Difference Between Preoperative and Postoperative QuickDASH Scores
Description: As assessed by the QuickDASH score, a patient reported outcome scale regarding hand disability. Higher scores indicate a patient's worse disability. This is to measure the difference in patient's disability before vs after their surgery.
Time Frame: One month postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale, 0 - 100
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
Number analyzed (Participants) | 17 | 17
score on a scale, 0 - 100 | 4.3 [-11.4 to 16.9] | 7.9 [-5.0 to 24.9]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the start of the study; i.e. patient's surgery, until the time of a patient's PACU discharge. This timeframe typically encompasses 1-3 hours, all on the same day.
Arm/Group | Usual Anesthesia Care | Virtual Reality Immersive Relaxation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT03614325/Prot_SAP_000.pdf